CLINICAL TRIAL: NCT04501029
Title: A Phase Ib/II Study of Gimatecan (ST1481) for Small Cell Lung Cancer Patients Who Failed Standard Platinum-containing Chemotherapy
Brief Title: A Study of Gimatecan (ST1481) in Small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Lee's Pharmaceutical Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ST1481-LEES-2020-03
Record Dates: First submitted 2020-07-30; First posted 2020-08-06 (Actual); Last update posted 2020-08-06 (Actual); Status verified 2020-07

CONDITIONS: Small Cell Lung Cancer
Keywords: small cell lung cancer; chemotherapy; gimatecan
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — ST 1481

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gimatecan group (Experimental): In Phase Ib study, patients will receive gimatecan at different dose level (0.4mg/m2, 0.6mg/m2,0.8mg/m2, oral, every 4 weeks) until progressive disease (PD).In Phase II study, patients will receive gimatecan at recommended phase II dose level.
  Interventions: Drug: Gimatecan

INTERVENTIONS:
Drug: Gimatecan — Patients will receive gimatecan orally at the recommended dose level on day 1-5 every 4 weeks.
  Other Names: ST1481

SUMMARY:
This phase Ib/II clinical trial studies the safety and effect of Gimatecan in small cell lung cancer patients who failed the first-line standard platinum-containing chemotherapy. The chemotherapy will be given every four weeks.

ELIGIBILITY:
Key Inclusion Criteria:

1. Aged 18 to 75 years old of either gender;
2. A histopathological or cytological diagnosis of small cell lung cancer(SCLC);
3. Recurrence or progression disease after firstline platinum-containing chemotherapy and patients intolerant or unwilling to receive standard treatment;
4. Measurable cancer lesion according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1;
5. Eastern Cooperative Oncology Group(ECOG) performance status score 0-1;
6. Estimated life expectancy >4 months;
7. Taking drugs orally;
8. The function of important organs meets the following requirements:

   1. white blood cell count (WBC) ≥ 4.0×109/L, absolute neutrophil count (ANC) ≥ 1.5×109/L, platelets ≥ 100×109/L, hemoglobin ≥ 90g/L;
   2. ALT, AST and AKP ≤ 2.5×ULN; liver metastasis: ALT、AST≤ 5.0×ULN, ALP ≤ 6.0×ULN; bone metastases ALT、AST≤ 2.5×ULN, ALP ≤ 5.0×ULN;
   3. serum albumin ≥ 30g/L;
   4. total bilirubin ≤ 1.5×ULN;
   5. serum creatinine ≤ 1.5×ULN, creatinine clearance rate ≥60 mL/min;
   6. INR ≤ 1.5, PT≤ 1.5×ULN;

10. Serum HCG negative in premenopausal women, female patients of childbearing potential and male patients with female partners of childbearing potential must be willing to avoid pregnancy; 11. Ability to understand the study and sign informed consent.

Key exclusion Criteria:

1. Patients who have been treated previously for SCLC with two system chemotherapy (except for targeted therapy, immunotherapy and antiangiogenic therapy);
2. Patients who have been treated previously with topotecan, Irinotecan or other topoisomerase I inhibitors;
3. Known or suspected allergy or hypersensitivity to the investigational drug gimatecan ingredients or their analogues;
4. Other anticancer therapy including any investigational agent within 28 days prior to the first dose of the investigational drug gimatecan;
5. Patients who have been treated previously with intravenous or oral drugs that affect CYP isoenzymes within 7 days prior to the first dose of the investigational drug gimatecan;
6. Brain metastasis or meningeal metastasis (except for asymptomatic patients with lesion stable more than 28 days);
7. Major surgical intervention or trauma within 28 days prior to the first dose of investigational drug administration;
8. A history of gastrointestinal disease which affects drug absorption;
9. A history of allogeneic stem cell transplantation and organ transplantation;
10. A history of interstitial lung disease or non-infectious pneumonia;
11. Patients who cannot tolerate chemotherapy due to severe cardiac, lung, liver or kidney dysfunction, or hematopoietic disease or cachexia;
12. A history of immunodeficiency (including a positive HIV test result), or other acquired or congenital immunodeficiency diseases;
13. Presence of active hepatitis B (HBV DNA ≥ 200 IU/mL or 103 copies/mL), hepatitis C (positive for hepatitis C antibody, and HCV-RNA levels higher than the lower limit of the assay);
14. A history of active pulmonary tuberculosis infection within 1 year or a history of active pulmonary tuberculosis infection more than 1 year ago but without formal anti-tuberculosis treatment;
15. A history of malignancies other than esophageal cancer before enrollment, excluding non-melanoma skin cancer, in situ cervical cancer, or cured early prostate cancer;
16. Pregnant or lactating women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2022-10-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
Dose limited toxicity (DLT) | up to 28 days.
  Phase Ib: Number of patients experienced any dose limited toxicity over the DLT period.
Recommended phase II dose (RP2D) | up to 12 months.
  Phase Ib: Determination of recommended phase II dose of escalating dose of gimatecan for the phase II part of the study.
Objective response rate (ORR) | To evaluate objective response rate every 8 weeks after the initiation of chemotherapy, up to 24 months.
  Percentage of patients with objective response assessed by best overall response (BOR) of either complete response(CR) or partial remission(PR) will be reported.

SECONDARY OUTCOMES:
Progression free survival (PFS) | From date of randomization until the date of death from any cause or the date of first documented disease progression whichever came first, assessed up to 24 months.
  The 2-year progression free survival of the whole group.
Disease control rate (DCR) | To evaluate disease control rate every 8 weeks after the initiation of chemotherapy, up to 24 months.
  Percentage of patients with disease control as assessed by best overall response (BOR) of either complete response(CR), partial remission(PR) or stable disease (SD) will be reported.
Duration of Response (DoR) | First documented CR or PR, whichever is first recorded until the first assessment of PD, assessed up to 24 months.
  The DoR applies only to patients whose BOR is either CR or PR. The duration is measured from the first documented response (CR or PR, whichever is first recorded) until the first assessment of Progressive Disease (PD).
Overall survival (OS) | From date of randomization until the date of death from any cause or the date of last follow-up whichever came first, assessed up to 24 months.
  The 2-year overall survival of the whole group.
Survival rate (SR) | up to 24 months.
  Survival probability of patients calculated according to Kaplan-Meier curve at either 1 or 2 year.
Treatment related adverse events rate | From the enrollment to 30 days later of the last chemotherapy.
  The incidence rate of treatment related adverse events of the whole group assessed by CTCAE v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: LIU XIAOQING, MD, Study Director — The Fifth Medical Center of the Chinese PLA General Hospital
Locations (1):
- The Fifth Medical Center of General Hospital of the Chinese People's Liberation Army, Beijing, Beijing Municipality, China

REFERENCES:
- [Result] Hurwitz JL, McCoy F, Scullin P, Fennell DA. New advances in the second-line treatment of small cell lung cancer. Oncologist. 2009 Oct;14(10):986-94. doi: 10.1634/theoncologist.2009-0026. Epub 2009 Oct 9. PMID 19819917
- [Result] Owonikoko TK, Behera M, Chen Z, Bhimani C, Curran WJ, Khuri FR, Ramalingam SS. A systematic analysis of efficacy of second-line chemotherapy in sensitive and refractory small-cell lung cancer. J Thorac Oncol. 2012 May;7(5):866-72. doi: 10.1097/JTO.0b013e31824c7f4b. PMID 22722788